CLINICAL TRIAL: NCT04354519
Title: The UK MS Regsiter COVID-19 Substudy
Brief Title: The United Kingdom Multiple Sclerosis Register Covid-19 Substudy
Acronym: UKMSRCV19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Swansea University (Other)
Responsible Party: Sponsor
Other Study IDs: 16SW0194
Record Dates: First submitted 2020-04-06; First posted 2020-04-21 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-05

CONDITIONS: Multiple Sclerosis; COVID-19
MeSH Terms: conditions — Multiple Sclerosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Confirmed Cases: Diagnosed by health professional / Covid-19 test
  Monitored through fortnightly questionnaires
- Not Covid-19 cases: Through self report no suspicion of COVID-19, tested by fortnightly questionnaire.
  non Covid Cases can become COVID cases through self report.
- Suspected Covid-19 Cases: Participants that are suspected of having Covid-19 but this has not been confirmed by health professional or Covid-19 test has not been performed.
  Fortnighly questionnaire

SUMMARY:
The aim of the study is to understand the impact of COVID-19 on People with Multiple Sclerosis in the United Kingdom.

DETAILED DESCRIPTION:
Study objectives

1. To identify the incidence of upper respiratory tract symptoms: fever, cough and breathing difficulties, other symptoms suggestive of COVID-19 infection, respiratory tract infections suggestive of COVID-19, and COVID-19 confirmed by laboratory testing among the UK MS population
2. To establish if some DMDs increase the risk of COVID-19 infection
3. To determine the incidence and effectiveness of self-isolation in the MS population. To examine the impact self-isolation has on mood, fatigue, and other routinely collected patient reported outcome measures from the MS Register.
4. To determine the clinical outcome of respiratory tract infections, including confirmed and suspected cases of COVID-19, in terms of symptoms, time to recovery, hospital admission, requirement for ventilation, and death.
5. To determine the longer-term impact of COVID-19 on MS, using routinely collected MS outcomes in the MS register, including impact on disability, relapses and changes in DMDs as assessed at 3 monthly intervals.
6. To determine where people are obtaining their health information during the COVID-19 outbreak.
7. To establish changes in DMDs prior to and as a result of symptoms related and unrelated to COVID-19

ELIGIBILITY:
Inclusion Criteria:

* >18 and confirmed diagnosis of MS, enrolled on UK MS Register

Exclusion Criteria:

* None of the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PwMS in the UK who self report as having MS, or have been recruited at a clinical site.
  Given the potentially vulnerable nature of pwMS due to active drug treatment and their potential susceptibility to infection it is important to chart this population within the MS Register
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-03-14 (Actual); Primary Completion 2022-07-14 (Estimated); Study Completion 2022-07-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of COVID-19 Infections within an MS Cohort in the UK | Through study completion, an average of 1 year
  Targeted questionnaire dependent on COVID Status
Hospitalisations in MS Patients with COVID-19 | 1 Year (regular outputs)
  Monitor admission rates in linked population
Mortality | 1 Year from study commencement
  Death data from routinely reported government level data (HES/PEDW)

SECONDARY OUTCOMES:
Patient Reported Expanded Disability Status Score | 1 year (at least 6 monthly)
  Patient Reported Outcome for MS disability
Hospital Anxiety and Depression Scale | 1 year (at least 6 monthly)
  Patient Reported Outcome for anxiety and depression
Multiple Sclerosis Impact Scale 29 V2 | 1 year (at least 6 monthly)
  Patient Reported Outcome for Multiple sclerosis impact on physical and psychological status
Multiple Sclerosis Walking Scale 12 V2 | 1 year (at least 6 monthly)
  Patient Reported Outcome for walking status
Fatigue Severity Scale | 1 year (at least 6 monthly)
  Patient Reported Outcome for impact of fatigue
EuroQol 5D (3l) | 1 year (at least 6 monthly)
  Patient Reported Outcome for general quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Nicholas, Principal Investigator — Clinical Lead; Nikos Evangelou, Principal Investigator — Co-PI
Locations (1):
- Swansea Univeristy, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Aggregate results will be published Line level data avaialble to other Researchers subject to Governance approval within Secure e-Research Platform

REFERENCES:
- See also: Main study website — https://ukmsregister.org/
- See also: Blog on the planned study — https://multiple-sclerosis-research.org/2020/03/guest-post-dr-richard-nicholas/

DOCUMENTS (1):
  • Study Protocol (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT04354519/Prot_000.pdf